CLINICAL TRIAL: NCT06523764
Title: Efficacy and Safety of Tegoprazan and Minocycline Dual Therapy for Helicobacter Pylori Initial Treatment : A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Tegoprazan and Minocycline Dual Therapy for Helicobacter Pylori Initial Treatment
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20242230-C-1
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Helicobacter Pylori Infection Chronic Gastrit
MeSH Terms: interventions — tegoprazan; Minocycline; Esomeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tegoprazan and minocycline dual theropy (Experimental): tegoprazan 50 mg and minocycline 100 mg by mouth, twice daily for 14 days
  Interventions: Drug: tegoprazan; Drug: Minocycline
- Bismuth-containing quadruple therapy (Active Comparator): bismuth potassium citrate 240 mg,esomeprazole 40 mg, amoxicillin 1000mg, and clarithromycin 500 mg by mouth,twice daily for 14 days
  Interventions: Drug: bismuth potassium citrate; Drug: Esomeprazole 40mg; Drug: Amoxicillin; Drug: clarithromycin

INTERVENTIONS:
Drug: tegoprazan — tegoprazan 50 mg and minocycline 100 mg by mouth, twice daily for 14 days
  Other Names: minocycline
  Arms: tegoprazan and minocycline dual theropy
Drug: Minocycline — tegoprazan 50 mg and minocycline 100 mg by mouth, twice daily for 14 days
  Arms: tegoprazan and minocycline dual theropy
Drug: bismuth potassium citrate — bismuth potassium citrate 240 mg,esomeprazole 40 mg, amoxicillin 1000mg, and clarithromycin 500 mg by mouth,twice daily for 14 days
  Arms: Bismuth-containing quadruple therapy
Drug: Esomeprazole 40mg — bismuth potassium citrate 240 mg,esomeprazole 40 mg, amoxicillin 1000mg, and clarithromycin 500 mg by mouth,twice daily for 14 days
  Arms: Bismuth-containing quadruple therapy
Drug: Amoxicillin — bismuth potassium citrate 240 mg,esomeprazole 40 mg, amoxicillin 1000mg, and clarithromycin 500 mg by mouth,twice daily for 14 days
  Arms: Bismuth-containing quadruple therapy
Drug: clarithromycin — bismuth potassium citrate 240 mg,esomeprazole 40 mg, amoxicillin 1000mg, and clarithromycin 500 mg by mouth,twice daily for 14 days
  Arms: Bismuth-containing quadruple therapy

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of tegoprazan and minocycline dual therapy for Helicobacter pylori initial treatment. It is hypothesized that tegoprazan and minocycline dual therapy is non-inferior to bismuth-containing quadruple therapy.Patients diagnosed with H. pylori infection will be randomly divided into one of the above treatments. At week 6 follow-up visits, a urea breath test#rapid urease test or helicobacter pylori stool antigen test will be performed to confirm eradication.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~70,both gender.
2. Patients with documented H.pylori infection who did not receive Helicobacter pylori eradication treatment;
3. Patients are willing to receive eradication treatment.
4. Women of childbearing age were required to use medically acceptable contraceptive methods during and 30 days after th

Exclusion Criteria:

1. Patients with contraindications or allergies to the study drug.
2. Severe organ damage and complications (such as liver cirrhosis, uremia, etc.), severe or unstable cardiopulmonary or endocrine diseases.
3. Constant use of anti-ulcer drugs ( including taking proton- pump.inhibitors(PPI) within 2 weeks before the [13C] urea breath test),antibiotics or bismuth complexes (more than 3 times /1 month before screening).
4. Pregnant or lactating women.
5. Underwent upper gastrointestinal Surgery.
6. Patients with moderate to severe dysplasia or high degree of intraepithelial neopla
7. Patients have symptom of dysphagia.
8. Evidence of bleeding or iron efficiency anemia.
9. A history of malignancy.
10. Drug or alcohol abuse history in the past 1 year.
11. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs,anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
12. Patients who has psychological problem or poor compliance.
13. Enrolled in other clinical trials in the past 3 months.
14. Refuse to sign informed conse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | 28 days after treatment
  The primary end point of this study is H.pylori eradication,established by negative urea breath test#rapid urease test or helicobacter pylori stool antigen test 28 days after the end of treament

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety) | 14 days of treatment
  Newly occurring drug-related symptoms during the treatment process
Rate of participants with good medication compliance (Compliance) | 14 days of treatment
  Taking more than 80% of medication is defined as good compliance

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi,, Principal Investigator — Chinaa, Shaanxi Xijing Hosipital of Digestive Disease
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No